CLINICAL TRIAL: NCT03273842
Title: Phase 1, Randomized Open Label, Multiple Dose, Parallel Study To Assess The Immunogenicity Of Multiple Subcutaneous (SC) Doses Of The Proposed Pegfilgrastim Biosimilar (PF-06881894) And Us-approved Neulasta (Registered) In Healthy Volunteers
Brief Title: A Study to Assess Immune Response to Multiple Doses of PF-06881894 or US-Approved Neulasta in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C1221005; IMM HSP-130 (Other: Alias Study Number)
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06881894 (Experimental): PF-06881894 6 mg SC
  Interventions: Biological: PF-06881894
- US-approved Neulasta (Active Comparator): US-approved Neulasta 6 mg SC
  Interventions: Biological: US-approved Neulasta

INTERVENTIONS:
Biological: PF-06881894 — pre-filled syringe 6 mg
  Arms: PF-06881894
Biological: US-approved Neulasta — pre-filled syringe 6 mg
  Arms: US-approved Neulasta

SUMMARY:
This study compares the immune response to the proposed biosimilar PF-06881894 and the US-approved Neulasta reference product. Subjects will receive 2 subcutaneous injections (6 milligrams [mg]) either 1 of the 2 study drugs. Subjects will receive the first dose on Day 1 of Period 1 and the second dose on Day 1 of Period 2. Pre-dose and serial post-dose assessments of immunogenicity will be conducted each of the two treatment periods. In addition, safety assessments will be conducted throughout the study.

ELIGIBILITY:
Inclusion Criteria:

• Healthy males or females between 18 and 65 years of age (both inclusive) with body mass index between 19 and 30 kg/m2, inclusive, and body weight of not <50 kg or >95 kg, will be enrolled in this study.

Exclusion Criteria:

* Hematologic laboratory abnormalities (including leukocytosis [defined as total leukocytes >11,000/mcL], leukopenia [defined as total leukocytes <4000/mcL], or neutropenia [defined as absolute neutrophil count <1500/mcL] or thrombocytopenia [defined as platelet count of <150,000/mcL]) or other clinically significant abnormal laboratory evaluations.
* Lack of adequate hepatic or renal reserve.
* Any active systemic or immunologic disease or condition.
* History of biological growth factor exposure.
* Received live vaccination or exposure to communicable viral diseases within 4 weeks prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with a negative baseline anti-pegfilgrastim antibody test result and confirmed postdose positive anti-pegfilgrastim antibody test result at any time during the study. | 90 days (through Period 1 Day1 to Period 2 Day 60 or final visit)

SECONDARY OUTCOMES:
The proportion of subjects with a negative baseline anti-pegfilgrastim antibody test result and postdose positive neutralizing antibody result at any time during the study. | 90 Days (through Period 1 Day 1 to Period 2 Day 60 or final study visit)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Seaview A Quotient Clinical Business, Coral Gables, Florida
  - Quotient Sciences- Jacksonville, LLC, Jacksonville, Florida
  - Seaview A Quotient Clinical Business, Miami, Florida
  - Vince & Associates Clinical Research Inc., Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Moosavi S, Borema T, Ewesuedo R, Harris S, Levy J, May TB, Summers M, Thomas JS, Zhang J, Yao HM. PF-06881894, a Proposed Biosimilar to Pegfilgrastim, Versus US-Licensed and EU-Approved Pegfilgrastim Reference Products (Neulasta(R)): Pharmacodynamics, Pharmacokinetics, Immunogenicity, and Safety of Single or Multiple Subcutaneous Doses in Healthy Volunteers. Adv Ther. 2020 Jul;37(7):3370-3391. doi: 10.1007/s12325-020-01387-x. Epub 2020 Jun 10. PMID 32524499
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1221005&StudyName=Phase+1%2C+Randomized+Open+Label%2C+Multiple+Dose%2C+Parallel+Study+To+Assess+The+Immunogenicity+Of+Multiple+Subcutaneous+%28sc%29+Doses+Of+The+Proposed+Pegfilgrastim+Biosimilar+%28pf-06881894%29+And+Us-approved+Neulasta+%28registered%29+In+Healthy+Volunteers